CLINICAL TRIAL: NCT00427973
Title: A Phase II Study of AZD2171 in Hepatocellular Carcinoma
Brief Title: AZD2171 in Treating Patients With Locally Advanced Unresectable or Metastatic Liver Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped prior to 2nd stage.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00130; 05-311 (Other: DFHCC IRB); N02CO12400 (Other Grant/Funding Number: US NIH Grant/Contract Award Number); CDR0000526405 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AZD2171 (Experimental): Patients will receive AZD2171 (cediranib maleate) 30mg by mouth once a day. Treatment may continue for as long as benefit is shown. Patients will undergo MRI and CT scan of the liver before beginning treatment, 3 days after the first dose of AZD2171, and after finishing course one. Patients will also undergo blood collection periodically for laboratory studies. Laboratory biomarker analysis, computed tomography, dynamic contrast-enhanced magnetic resonance imaging, and pharmacological study will be performed.
  Interventions: Drug: cediranib maleate; Other: laboratory biomarker analysis; Procedure: computed tomography; Procedure: dynamic contrast-enhanced magnetic resonance imaging; Other: pharmacological study

INTERVENTIONS:
Drug: cediranib maleate — Given orally
  Other Names: AZD2171
Other: laboratory biomarker analysis — Peripheral blood was obtained from all patients enrolled for studies of early changes in circulating proangiogenic and proinflammatory molecules and cells. Blood samples were collected in EDTA-containing tubes before and after cediranib therapy on days 1 and 14 of cycle 1. Circulating VEGF, placental growth factor (PlGF), sVEGFR1, basic fibroblast growth factor (bFGF), interleukin (IL)-6, IL-8, transforming growth factor a ((TNF-a), gamma interferon (IFN-g) were measured using multiplex ELISA plates from Meso-Scale Discovery. Hepatocyte growth factor (HGF), insulin-like growth factor 1 (IGF-1), sVEGFR2, angiopoietin 2 (Ang-2), sTie2, soluble c-KIT, carbon anhydrase 9 (CAIX), and stromal cell-derived factor-1a (SDF1a) were measured using ELISA kits from R&D Systems.
Procedure: computed tomography — computed tomography (CT) every 8 weeks to evaluate response and progression.
Procedure: dynamic contrast-enhanced magnetic resonance imaging — Magnetic resonance imaging (MRI) every 8 weeks to evaluate response and progression.
  Other Names: DCE-MRI
Other: pharmacological study — Blood samples to characterize the steady-state PK of cediranib were drawn from a peripheral vein shortly before patients received the dose on days 8 and 15 of cycle 1 and at the following times relative to dosing on day 1 of cycle 2: 5 min and 1, 2, 4, 6, 8, and 24 hours, with the last sample collected before taking the next daily dose.
  Other Names: pharmacological studies

SUMMARY:
This phase II trial is studying how well AZD2171 works in treating patients with locally advanced unresectable or metastatic liver cancer. AZD2171 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the progression free survival of patients with locally advanced unresectable or metastatic hepatocellular carcinoma treated with AZD2171.

SECONDARY OBJECTIVES:

I. Determine the toxicity of this drug in these patients. II. Determine, preliminarily, the efficacy of this drug, in terms of response rate, duration of response, and overall survival, in these patients.

III. Determine the blood flow changes and vascular permeability of the tumor in patients treated with this drug.

IV. Determine the pharmacokinetic profile of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral AZD2171 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Dynamic contrast-enhanced (DCE) MRI and CT perfusion scan of the liver are performed at baseline, 72 hours after the initial dose of AZD2171, and at the end of course 1. Blood samples for pharmacokinetic studies are collected periodically during study.

After the completion of study treatment, patients are followed every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed hepatocellular carcinoma
* Locally advanced unresectable OR metastatic disease
* Cancer of the Liver Italian Program (CLIP) score =< 3
* Symptomatic congestive heart failure
* Unstable angina pectoris
* Measurable disease, defined as >= 1 unidimensionally measurable lesion>= 20 mm by conventional techniques OR >= 10 mm by spiral CT scan
* Cardiac arrhythmia
* Measurable lesion must be outside field of prior chemoembolization
* No known brain metastases
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* Absolute neutrophil count >= 1,000/mm^3
* Platelet count >= 75,000/mm^3
* Hemoglobin >= 8 g/dL
* Bilirubin =< 3.0 mg/dL
* AST and ALT =< 7 times upper limit of normal
* Creatinine =< 2.0 mg/dL
* Fertile patients must use effective contraception
* CLIP score =< 3

Exclusion Criteria:

* Not pregnant or nursing
* Negative pregnancy test
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to AZD2171
* No chronic diarrhea or any disorder that would limit adequate absorption of AZD2171
* No familial history of long QT syndrome
* Proteinuria =< +1 on two consecutive dipsticks taken no less than 1 week apart
* No other uncontrolled illness including, but not limited to, any of the following:
* Hypertension
* Ongoing or active infection
* No psychiatric illness or social situation that would limit study compliance
* Recovered from prior therapy
* Prior systemic chemotherapy regimens for hepatocellular carcinoma allowed
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* More than 4 weeks since prior radiotherapy, major surgery, or chemoembolization
* At least 30 days since prior participation in an investigational trial
* No other concurrent investigational agents
* No concurrent medication that may markedly affect renal function (e.g., vancomycin, amphotericin, or pentamidine)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer agents or therapies
* No mean QTc > 470 msec (with Bazett's correction) on screening EKG (490 msec for women)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-05; Primary Completion 2010-04 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zhu, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Zhu AX, Ancukiewicz M, Supko JG, Sahani DV, Blaszkowsky LS, Meyerhardt JA, Abrams TA, McCleary NJ, Bhargava P, Muzikansky A, Sheehan S, Regan E, Vasudev E, Knowles M, Fuchs CS, Ryan DP, Jain RK, Duda DG. Efficacy, safety, pharmacokinetics, and biomarkers of cediranib monotherapy in advanced hepatocellular carcinoma: a phase II study. Clin Cancer Res. 2013 Mar 15;19(6):1557-66. doi: 10.1158/1078-0432.CCR-12-3041. Epub 2013 Jan 29. PMID 23362324
- See also: pubmed article — http://www.ncbi.nlm.nih.gov/pubmed/23362324

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled the targeted 17 patients for the first stage between May 2009 and January 2010. Patients were recruited in the outpatient clinics.
Groups:
- Singe Arm Open Label Study With AZD2171 at 30 mg Daily.: Patients will receive AZD2171 by mouth once a day. Treatment may continue for as long as benefit is shown. Patients will undergo MRI and CT scan of the liver before beginning treatment, 3 days after the first dose of AZD2171, and after finishing course one. Patients will also undergo blood collection periodically for laboratory studies.
Period: Overall Study
Arm/Group | Singe Arm Open Label Study With AZD2171 at 30 mg Daily.
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Singe Arm Open Label Study With AZD2171 at 30 mg Daily: Patients will receive AZD2171 (cediranib maleate) by mouth once a day. Treatment may continue for as long as benefit is shown. Patients will undergo MRI and CT scan of the liver before beginning treatment, 3 days after the first dose of AZD2171, and after finishing course one. Patients will also undergo blood collection periodically for laboratory studies. Laboratory biomarker analysis, computed tomography, dynamic contrast-enhanced magnetic resonance imaging, and pharmacological study will be performed.
  cediranib maleate: Given orally
  laboratory biomarker analysis
  computed tomography
  dynamic contrast-enhanced magnetic resonance imaging
  pharmacological study
Arm/Group | Singe Arm Open Label Study With AZD2171 at 30 mg Daily
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: years] | 66 [46 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 17
Eastern Cooperative Oncology Group [Median (Full Range); unit: units on a scale] — Grade ECOG 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  units on a scale | 1 [0 to 2]
Cancer Of Liver Italian Program (CLIP) [Median (Full Range); unit: units on a scale] — CLIP score calculated by assigning a score (0, 1 or 2) to each of 4 clinical factors and then adding the 4 scores to arrive at the CLIP score. Higher values in each of the 4 clinical factors represent a worse outcome. CLIP score range (0-6) w/ higher values=worse outcome
  1. Child-Pugh:A=0, B=1, or C=2
  2. If tumor morphology is uninodal w/ extension <=50%, score=0, if multinodular and extension <=50%, score=1, if tumor morphology massive or extension >50%, score=2.
  3. AFP <400, score=0, AFP >=400, score=1.
  4. No portal vein thrombosis, score=0, portal vein thrombosis present, score=1.
  units on a scale | 2 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression is defined as a 20% increase in the sum of the of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions by conventional RECIST based criteria, or death, which ever comes first.
  This design yields at least 90% power to detect a true 3-month PFS rate of at least 69%.
Time Frame: 3 months
Population: The number of patients who were progression free at 3 months was determined. 13 of 17 patients (77%) were progression free at 3 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Singe Arm Open Label Study With AZD2171 at 30 mg Daily
Number analyzed (Participants) | 17
percentage of participants | 77 [60 to 99]

2. Secondary Outcome: Response Rate
Description: Number of patients who achieve either complete or partial response based on RECIST Criteria for target lesions assessed by MRI.
  Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 1 year
Population: Patients receiving AZD2171 (cediranib maleate)
Measure: Number; unit: participants with confirmed response
Arm/Group | Singe Arm Open Label Study With AZD2171 at 30 mg Daily
Number analyzed (Participants) | 17
participants with confirmed response | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival will be calculated using the Kaplan-Meier method, and confidence limits for survival estimates will be calculated using the Greenwood formula.
Time Frame: The time from study entry until death from any cause, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Singe Arm Open Label Study With AZD2171 at 30 mg Daily
Number analyzed (Participants) | 17
months | 11.7 [7.5 to 13.6]

4. Post Hoc Outcome: Discontinued Treatment Due to SAE
Description: Participants that discontinued treatment due to a Serious Adverse Event (SAE)
Time Frame: May 2009 through January 2010
Measure: Number; unit: Participants
Arm/Group | Singe Arm Open Label Study With AZD2171 at 30 mg Daily
Number analyzed (Participants) | 17
Participants | 0

ADVERSE EVENTS:
Description: A total of 77 treatment cycles were administered, with a median of 3 cycles per patient (range: 1-15). Twelve of 17 patients required dose interruptions and subsequent reductions for the following reasons: gr 3 elevated AST (3), gr 3 hyperbilirubinemia (3), gr 3 elevated ALT (2), gr 3 dehydration (1), gr 2 diarrhea (1), and gr 1 proteinuria (2).
Groups:
- Singe Arm Open Label Study With AZD2171 at 30 mg Daily: Patients will receive AZD2171 (cediranib maleate) at 30 mg by mouth once a day. Treatment may continue for as long as benefit is shown. Patients will undergo MRI and CT scan of the liver before beginning treatment, 3 days after the first dose of AZD2171, and after finishing course one. Patients will also undergo blood collection periodically for laboratory studies. Laboratory biomarker analysis, computed tomography, dynamic contrast-enhanced magnetic resonance imaging, and pharmacological study will be performed.
  cediranib maleate: Given orally
  laboratory biomarker analysis
  computed tomography
  dynamic contrast-enhanced magnetic resonance imaging
  pharmacological study
Arm/Group | Singe Arm Open Label Study With AZD2171 at 30 mg Daily
Serious Adverse Events (participants affected / at risk) | 5/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Singe Arm Open Label Study With AZD2171 at 30 mg Daily (N=17)
pulmonary embolism (Vascular disorders) | 1 (1)
hyperbilirubinemia (Gastrointestinal disorders) | 4 (4)
left subdural hemorrhage (Nervous system disorders) | 1 (1) — unwitnessed fall with mental status change and was found to have large left subdural hemorrhage and transtentorial herniation leading to death
Fatigue (General disorders) | 1 (1)
AST-SGOT (Gastrointestinal disorders) | 2 (2)
Hyponatremia (General disorders) | 5 (5)
Alk. Phosphatemia (Hepatobiliary disorders) | 1 (1)
ALT-SGPT (Gastrointestinal disorders) | 1 (1)
Hypertension (Cardiac disorders) | 5 (5)
Hypophosphatemia (General disorders) | 1 (1)
Proteinuria (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Cardiac Ischemia (Cardiac disorders) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Singe Arm Open Label Study With AZD2171 at 30 mg Daily (N=17)
Fatigue (General disorders) | 14 (14)
AST-SGOT (Gastrointestinal disorders) | 12 (12)
Hyponatremia (General disorders) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 10 (10)
Nausea (Immune system disorders) | 9 (9)
Alk.Phosphatemia (Hepatobiliary disorders) | 8 (8)
ALT-SGPT (Gastrointestinal disorders) | 8 (8)
Weight loss (General disorders) | 8 (8)
Anorexia (General disorders) | 7 (7)
Hyperbilirubinemia (Hepatobiliary disorders) | 7 (7)
Hypertension (Cardiac disorders) | 7 (7)
Hypophosphatemia (General disorders) | 7 (7)
Proteinuria (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (5)
Leukopenia (Investigations) | 5 (5)
Lymphopenia (Investigations) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (4)
Fever w/o neutropenia (General disorders) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypothyroidism (Endocrine disorders) | 3 (3)
Confusion (Psychiatric disorders) | 2 (2)
Creatinine (Investigations) | 2 (2)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Taste disturbance (Gastrointestinal disorders) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cardiac ischemia (Cardiac disorders) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Epistaxis (Social circumstances) | 1 (1)

LIMITATIONS AND CAVEATS:
Despite reaching the prespecified goal for the first stage of the trial, the study was stopped and did not proceed to the second stage after reviewing the development program of cediranib by AstraZeneca for reasons unrelated to this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less